CLINICAL TRIAL: NCT06320431
Title: A Multicentre, Prospective, Randomized, Open Label, Blinded-endpoint Trial to Optimize the Use of Intravenous Tenecteplase in Participants With Acute Ischemic Stroke (ACT-GLOBAL THROMBOLYSIS (ACT WHEN-001) Within A Multi-faCtorial, mulTi-arm, Multi-staGe, Randomised, gLOBal Adaptive pLatform Trial for Stroke (ACT-GLOBAL) NCT06352632
Brief Title: ACT-GLOBAL THROMBOLYSIS (ACT-WHEN-001) Domain Within the ACT-GLOBAL Adaptive Platform Trial-NCT06352632
Acronym: ACT-WHEN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: The George Institute for Global Health, Australia (Other)
Responsible Party: Principal Investigator, Dr. Bijoy Menon, MD, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACT-WHEN-001
Record Dates: First submitted 2024-02-05; First posted 2024-03-20 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2024-09

CONDITIONS: Acute Ischemic Stroke AIS; Stroke Acute; Stroke, Acute, Stroke Ischemic
Keywords: Stroke; Thrombolysis; Platform; Tenecteplase; Endovascular thrombectomy; EVT; Domain
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Intervention Model Description: Randomization will be stratified by: (1) planned emergency endovascular thrombectomy (EVT) and (2) known use or history to suggest use of a standard-dose direct oral anticoagulant (DOAC) within the last 48 hours. Randomization will be centralized, secure and concealed, using a web-based server and permuted blocks of varying sizes will be used.
  This will result in four pre-defined strata: (i) EVT+ / DOAC+ (ii) EVT+ / DOAC- (iii) EVT- / DOAC+ and (iv) EVT- / DOAC-.
  Patients in strata 1, 2 and 3 will be randomized to standard-dose IV tenecteplase (0.25 mg/kg body weight) vs. Low-dose tenecteplase (0.18 mg/kg body weight) or no IV thrombolysis (1:1:1 randomization). Patients in strata 4 will be randomized to standard-dose intravenous (IV) tenecteplase (0.25 mg/kg body weight) vs. Low-dose IV tenecteplase (0.18 mg/kg body weight) only (1:1 randomization).
  Emergency EVT is defined as anticipated arterial puncture time in the enrolling hospital ≤ 60 minutes from randomization.
Who Masked: Outcomes Assessor
Masking Description: The trial will have allocation concealment and blinded endpoint assessment, but open-label treatment. Given the time sensitive nature of acute stroke treatment, blinding the enrolling personnel to treatment assignment is not practical. Clinical site staff, including the Principal Investigator (PI), sub-investigators, clinic site staff, and the Sponsor will not be blinded to treatment allocated or received. In the event of an emergency the PI will be already unblinded.
  The trial will have blinded endpoint assessment on Day 90, with central blinded assessors contacting the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard-dose intravenous tenecteplase (0.25 mg/kg body weight) (No Intervention): The intervention group will receive intravenous tenecteplase as a single bolus as per the standard manufacturers' instructions for use. The dose administered will be 0.25 mg/kg body weight (maximum dose 25 mg) over 10-20 seconds as soon as possible after randomization.
- 2) IVT with tenecteplase at low-dose: 0.18 mg/kg (Active Comparator): The intervention group will receive intravenous tenecteplase as a single bolus as per the standard manufacturers' instructions for use. The dose administered will be 0.18 mg/kg body weight (maximum dose 18 mg) over 10-20 seconds as soon as possible after randomization.
  Interventions: Drug: Tenecteplase
- 3) No IV thrombolysis [(only in those undergoing EVT or those on DOACs) (Active Comparator): No intravenous tenecteplase only applied to subjects on DOACs over the last 24 hours or those planned for emergency EVT
  Interventions: Drug: Tenecteplase

INTERVENTIONS:
Drug: Tenecteplase — Thrombolytic
  Other Names: TNKase; Metalyse
  Arms: 2) IVT with tenecteplase at low-dose: 0.18 mg/kg; 3) No IV thrombolysis [(only in those undergoing EVT or those on DOACs)

SUMMARY:
This domain has a prospective, randomized, controlled, open-label, parallel group with blinded endpoint assessment (PROBE) design. Up to 4,000 patients with presumed acute ischemic stroke (AIS) will be followed for 90 days (or until death, if prior to 90 days). The end of the trial is defined as the date that all participants have completed their Day 90 assessment.

This domain aim is to efficiently, reliably, and simultaneously, determine the comparative effectiveness of intravenous thrombolysis (IVT) using standard-dose intravenous tenecteplase (0.25 mg/kg body weight), vs. low-dose intravenous tenecteplase (0.18 mg/kg body weight) in all patients who present to hospital with acute ischemic stroke and are considered for intravenous thrombolysis. In addition, this domain also seeks to study standard-dose intravenous tenecteplase (0.25 mg/kg body weight), vs. low-dose intravenous tenecteplase (0.18 mg/kg body weight) vs. no TNK upfront with rescue IA TNK if necessary (in those eligible for emergency EVT) and no TNK upfront in those who have taken DOACs during the preceding 48 hours. This domain therefore seeks to generate more robust randomized evidence to guide clinicians in their decisions over the balance of risks and treatment with intravenous thrombolysis with tenecteplase wherever such evidence is currently insufficient.

This domain will currently evaluate four research questions in relation to the use of IVT with tenecteplase:

1. In patients with recent (48 hours) intake of a standard-dose direct oral anticoagulant (DOAC), how should IVT be used? - Use standard-dose (0.25 mg/kg body weight) or low-dose tenecteplase (0.18 mg/kg) or not at all.
2. In patients planned to be treated with endovascular thrombectomy, how should tenecteplase be used? -Treat with IV tenecteplase (standard- or low-dose) or not at all.
3. In any patient receiving IVT, what is the optimal dose of tenecteplase? - use standard-dose (0.25 mg/kg body weight) or low-dose tenecteplase (0.18 mg/kg).
4. To what extent is the treatment effect of standard- vs. low-dose tenecteplase modified by key patient characteristics, such as diabetes, prior antiplatelet therapy, renal failure, or frailty, old age or having a heavy burden of cerebral small vessel disease on brain imaging.

DETAILED DESCRIPTION:
Background and Rationale:

Tenecteplase has become the first choice of IVT for patients with AIS in hospitals around the world: its mechanisms of action are well characterized; the single bolus administration has important practical advantages over alteplase (0.9 mg/kg, max. 90 mg; with 10% of the dose given as a bolus followed by an infusion over 60 mins); trials indicate it has non-inferior efficacy as compared to alteplase, potential superiority among patients with large-vessel occlusion; and it is endorsed by national and international guidelines. While alteplase remains the only regulatory-approved IVT for the treatment of AIS in some countries with tenecteplase (0.25 mg/kg body weight) recently approved by the European Medical Agency, it is anticipated that this will continue to change over the next year. Current evidence indicates tenecteplase is as safe, and potentially more efficacious than alteplase in AIS.

Optimal tenecteplase dosing:

Doses of tenecteplase ranging from 0.1 to 0.4mg/kg were tested in clinical trials of acute stroke with a dose of tenecteplase 0.25 mg/kg body weight showing comparable efficacy to standard dose alteplase (0.9 mg/kg body weight). When compared to standard dose alteplase, the large ENCHANTED trial that enrolled 3000 patients suggested that 2/3rd standard dose alteplase has better safety, with similar efficacy rates but failed to show statistical non-inferiority. This lower dose of alteplase is used as standard care in many Asian countries. With results from the recently completed AcT trial showing similar efficacy and safety of tenecteplase (0.25 mg/kg body weight) vs. standard dose alteplase (0.9 mg/kg body weight), tenecteplase at 0.25 mg/kg body weight is becoming the new global standard for intravenous thrombolysis. Dosing studies with intravenous tenecteplase have however not tested efficacy and safety of low dose (2/3rd standard dose) tenecteplase, like in the ENCHANTED trial, in a broad population of acute stroke patients. A network meta-analysis of five clinical trials suggested better efficacy with intravenous tenecteplase at 0.25mg/kg with better safety at 0.1mg/kg, as compared to 0.4mg/kg, the only three doses on which such data is available. While the Canadian Stroke Best Practices, European Stroke Organization Guidelines and multiple national guidelines recommend an intravenous tenecteplase dose of 0.25mg/kg to a maximum of 25mg for acute stroke under 4.5 hours, there are certain scenarios where thrombolysis may carry a higher theoretical risk of hemorrhagic complications, warranting a more cautious approach with a lower dose tenecteplase (0.18 mg/kg). This lower dose of tenecteplase (midway between 0.25 mg/kg and 0.1 mg/kg and approximately 2/3rd standard dose tenecteplase) may potentially offer an optimal balance of efficacy and safety in many patient risk groups.

Recent ingestion of DOACs:

This is now one of the most frequent reasons why IVT is not administered, being present in ~6% of all patients presenting with AIS. The large prospective multi-site national Swiss Stroke Registry conducted in 2014-2019 indicates that of all patients with AIS and known atrial fibrillation (AF) who were potentially eligible for IVT, 466 (18%) were on a DOAC and 247 (9.5%) were on prior warfarin anticoagulation, and the number and age of patients, and indications for DOAC use, has rapidly increased over time. Separately, a recently published large international registry and a meta-analysis of other observational studies show that prior intake of DOACs within 48 hours of alteplase is not associated with an increased risk of ICH. No study until now, has compared IVT with tenecteplase standard-dose vs. low-dose tenecteplase vs. no tenecteplase in a randomized manner in these patients.

EVT eligibility:

EVT is the biggest advance in AIS treatment in the last decade, used in patients with target intracranial occlusions typically in proximal large-vessels of the cerebral circulation. Reperfusion rates as high as 90% are achieved in such patients, with the number-needed-to-treat to achieve improved outcomes being as low as 2.6. Reperfusion rates continue to improve with better technology, techniques, and operator experience. Conversely, data indicate lower rates of recanalization with IVT where there are large-vessel occlusions (a third of the EVT rates and at a later time), raising concerns over the utility of IVT in these patients. A meta-analysis of recent data concluded EVT alone is non-inferior to IVT with standard-dose alteplase followed by EVT; with the lower boundary of the 95% confidence interval (CI) being -2%;34 and rates of symptomatic intracerebral hemorrhage were 1% higher in patients offered IVT+EVT vs. EVT alone. The recent IRIS collaboration patient level meta-analysis did not however establish the non-inferiority of EVT alone compared with IVT (with alteplase) plus EVT in patients presenting directly at EVT centers. No study has compared IVT with tenecteplase before EVT vs. EVT alone (with rescue IA tenecteplase if EVT fails), nor of standard-dose vs. low-dose tenecteplase, in these patients. Our survey shows physicians persist in their uncertainty over how and when to use thrombolysis with tenecteplase in EVT-eligible patients.

The elderly, frail and those with comorbidities:

Age is one of the most important prognostic factors for outcomes in AIS. Multiple studies have shown that older age is associated with poor outcome and an increased risk of ICH with IVT. Underlying conditions such as renal failure, diabetes, cerebral small vessel disease, and remote cerebral infarcts, which increase the risks of ICH, are more frequently detected with modern brain imaging and are more common in the elderly. However, the elderly have often been excluded from acute stroke trials, such as in the original NINDS trial of alteplase where only 69 subjects over the age of 80 years were included, and similar figures in the subsequent ECASS III trial that sought to establish the efficacy of IVT in the 3-4.5-hour time window. Most of the randomized data for IVT in this age group have come from the IST-3 trial, which included 1,711 elderly patients; the rest of the data on the effectiveness of IVT in the elderly comes from registry studies (e.g. SITS, VISTA and SPOTRIAS), all on alteplase. In the ENCHANTED and AcT trials, there was no significant heterogeneity in the treatment effect by age. Although guidelines recommend the use of IVT in the elderly, they qualify this with caution over the risks of ICH and assign lower grades of evidence on efficacy in patients presenting late from symptom onset. A lower dose of tenecteplase could offer a safer and potentially more effective strategy in the elderly with AIS.

Patients with sub-acute looking infarcts, small intraarterial thrombi or no visible occlusions on baseline imaging:

Modern stroke imaging techniques are better able to characterize risk of ICH with IVT as compared to clinical judgement alone. Sub-acute looking infarcts (regions of the brain with moderate to severe hypoattenuation on non-contrast CT) can be seen early after stroke onset and signify severe ischemia. They are associated with higher risk of ICH; other studies show that benefit of IVT remains even with this higher ICH risk. Patients with small intra-arterial thrombi recanalize better with IVT than those with larger thrombi. In the ENCHANTED trial, patients with small or no visible occlusions on CT Angiography did better with low-dose vs. standard-dose alteplase. In subgroup analyses of the IST-3 trial, patients with no visible occlusions on baseline CT or MR angiography fared worst with standard-dose alteplase than when treated conservatively. There are no studies that assess risks and benefits of thrombolysis with tenecteplase (standard vs. low dose tenecteplase) when imaging assessed risks are potentially high or when thrombus burden itself is low.

Patients with dementia:

Although dementia itself is not a contraindication for IVT in patients presenting with acute ischemic stroke, these patients have not been included in most clinical trials on thrombolysis because dementia may confound neurological assessments, or their prognosis is so poor that discriminating a treatment effect would not be possible. Moreover, common conditions causally related to dementia include previous strokes and microbleeds associated with amyloid angiopathy, thus raising concerns about risk of ICH with thrombolysis. A propensity score matched analysis of data from the registry of the Canadian Stroke Network showed no differences between those with and without dementia in the risk of intracerebral hemorrhage, in mortality or in disability at discharge when administered IVT. In the Nationwide Inpatient Sample study however, dementia was associated with increased risk of symptomatic ICH in patients administered IVT. Randomized data on optimal dose of IVT with tenecteplase, especially in the context of pre-existing dementia/cognitive impairment is lacking.

Other patient groups:

There are many other patient groups where evidence gaps exist, guidelines offer some recommendations regarding IVT, but physicians continue to have uncertainties. These include those with high blood sugar or blood pressure at presentation, those with pre-existing severe renal dysfunction or those with functional disabilities. Some of these conditions are more prevalent than others; some patients have more than one of these conditions. With many of these patients, physician uncertainties vary around the degree/extent of these conditions and not just their presence or absence. Race and ethnic differences have also been noted with risk of ICH post IVT. Blacks and Asians likely have higher risk of ICH than Hispanics and Whites. Sex differences exist with women being offered less IVT (10% less than men in some studies) even after adjusting for all other variables.

Data from a large adaptive randomized clinical trial on thrombolysis dose and safety with tenecteplase, in the various patient conditions described above, will increase physician confidence and potentially result in better and faster utilization of intravenous thrombolysis, thus helping improve patient outcomes overall.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with disabling AIS presenting within 4.5 hours of symptom onset or last known well who may benefit from intravenous thrombolysis (IVT) with tenecteplase. Patients potentially eligible for IVT with conditions described as relative contraindications in national guidelines where physician discretion is recommended are eligible. Patients who received a DOAC, and those planned for emergency EVT are eligible.
2. Consent process completed as per national laws and regulation and the applicable ethics committee requirements.

Exclusion Criteria:

1. Any absolute contraindication for IV thrombolysis per current national guidelines. Examples include those who are actively bleeding, had recent intracranial surgery, head trauma, intracranial or subarachnoid hemorrhage, or a bleeding diathesis.
2. Minor stroke patients with non-disabling symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
A reduction of functional dependence analyzed across the whole distribution of outcomes assessed on the modified Rankin Scale (mRS), | From enrollment to the Day 90 assessment - Day 90 outcomes are assessed in a blinded manner
  Modified Rankin Scale (mRS) -which scores of 0 to 1 indicate a favourable outcome without or with symptoms but no disability, scores of 2 to 5 indicate increasing levels of disability (and dependency), and a score of 6 indicates death.

SECONDARY OUTCOMES:
90-day mortality | From enrollment to the Day 90 assessment.
  Date and cause of death are collected from randomization until End of Study.
Proportion of participants with a Modified Rankin Scale (mRS) of 0-1 at Day 90. | Completed by telephone at the Day 90 assessment (Day 90 outcomes are assessed in a blinded manner)
  Modified Rankin Scale (mRS) -which scores of 0 to 1 indicate a favourable outcome without or with symptoms but no disability, scores of 2 to 5 indicate increasing levels of disability (and dependency), and a score of 6 indicates death.
Proportion of participants with a Modified Rankin Scale (mRS) of 0-2 at Day 90. | Completed by telephone at the Day 90 assessment (Day 90 outcomes are assessed in a blinded manner)
  Modified Rankin Scale (mRS) -which scores of 0 to 1 indicate a favourable outcome without or with symptoms but no disability, scores of 2 to 5 indicate increasing levels of disability (and dependency), and a score of 6 indicates death.
Health-related quality of life, as measured by the EQ-5D-5L at Day 90. | Completed by telephone at the Day 90 assessment (Day 90 outcomes are assessed in a blinded manner)
  The EQ-5D-5L is a generic instrument for describing and valuing health. It is based on a descriptive system that defines health in terms of five dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has five response categories corresponding to: no problems, slight, moderate, severe and extreme problems. The version of the instrument selected for the trial is interviewer administered either in-person, or by telemedicine or by telephone. The respondents will also rate their overall health on the day of the interview on a 0-100 visual analogue scale (EQ-VAS).
The frequencies of Serious Adverse Events (SAEs) from enrollment up to Day 4 | From enrollment ( randomization) to the Day 4
  Serious Adverse events include the following events :results in death, life threatening,Requires inpatient hospitalization or prolongation of existing hospitalization,Results in persistent disability/incapacity,Is a congenital anomaly/birth defect, an important medical event that may not result in death, be life-threatening, or require hospitalization, but may jeopardize the participant and may require medical or surgical intervention to prevent an outcome listed in the SAE selection.
Symptomatic intracranial hemorrhage | Up to 36 hours from randomization
  Any new intracranial hemorrhage detected by brain imaging associated with neuroligical worsening or deterioration of symptoms.
Large parenchymal hemorrhage (PH-2) | up to 36 hours from randomization
  PH-2:( hemorrhage grading scale) homogeneous hyperdensity occupying over 30% of the infarct zone, with significant mass effect
Ordinal shift of 7 levels of mRS at 90 days | Done by telephone at the Day 90 assessment (Day 90 outcomes are assessed in a blinded manner)
  Modified Rankin Scale (mRS) -which scores of 0 to 1 indicate a favourable outcome without or with symptoms but no disability, scores of 2 to 5 indicate increasing levels of disability (and dependency), and a score of 6 indicates death.
Proportion of participants achieving first pass (eTICI 2c or higher) reperfusion (when treated with EVT). | Assessed and evaluated after the EVT procedure by the Central Imaging Core lab by blinded radiologists/stroke neurologists-the imaging reading will be done over the course of the trial through study completion.
  The thrombolysis in cerebral infarction (TICI) grading system was described in 2003 by Higashida et al. as a tool for determining the response of thrombolytic therapy for ischemic stroke. In neurointerventional radiology it is commonly used for patients post endovascular revascularization.
Proportion of participants achieving successful recanalization (revised arterial occlusive lesion [rAOL] score of 2b-3) at first angiographic acquisition (when treated with EVT). | Assessed and evaluated after the EVT procedure by the Central Imaging Core lab by blinded radiologists/stroke neurologists. These imaging readings will be done over the course of the trial through study completion.
  The thrombolysis in cerebral infarction (TICI) grading system was described in 2003 by Higashida et al. as a tool for determining the response of thrombolytic therapy for ischemic stroke. In neurointerventional radiology it is commonly used for patients post endovascular revascularization.
Ambulatory status at discharge | Completed the day the patient is discharged from hospital.
  Assessing mobility of the patient at discharge
Place of residence at 90 days | Completed at the Day 90 follow-up visit
  Assessing the patient's residence at the Day 90 follow up. ( example: home,rehabilitation, long term care, remains hospitalized)
Imaging assessment (e.g., infarct size and edema volume) | Assessed and evaluated by the Central Imaging Core lab by blinded radiologists/stroke neurologists. These imaging readings will be performed over the course of the trial through study completion.
  The total absolute infarct volume is the sum of infarct volumes calculated for each slice.
Summative total length of hospital stay in the first 90-days after stroke onset | Completed at the Day 90 follow-up visit.
  Calculating the total number of days the patient was hospitalized since their hospital admission.

CONTACTS AND LOCATIONS:
Overall Officials: Bijoy K Menon, MD, Principal Investigator — University of Calgary; Craig Anderson, MD, Principal Investigator — The George Institute
Locations (24):
- Australia (3):
  - The George Institute for Global Health, Sydney, Barangaroo
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Monash University (Box Hill), Melbourne, Victoria
- Canada (21):
  - University of Calgary, Calgary, Alberta
  - Medicine Hat Regional Hospital, Medicine Hat, Alberta
  - Red Deer Regional Hospital, Red Deer, Alberta
  - University of Alberta, Edmonton, A
  - Kelowna Regional Hospital, Kelowna, British Columbia
  - Royal Columbian Hospital, New Westminster, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - Brandon Regional Hospital, Brandon, Manitoba
  - University of Manitoba - Winnipeg Health Science Centre, Winnipeg, Manitoba
  - Queen Elizabeth II Health Science Center (Halifax), Halifax, Nova Scotia
  - Health Sciences North Horizon Sante-Nord, Greater Sudbury, Ontario
  - McMaster University Hamilton Health Sciences Centre, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Lawson Health Research Institute- London, London, Ontario
  - University of Ottawa, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Queen Elizabeth Hospital (PEI), Charlottetown, Prince Edward Island
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS Fleurimont Hôpital (Sherbrooke), Sherbrooke, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No
Domain information and tabular trial results will be posted on the National Institutes of Health's website www.clinicaltrials.gov within one year of domain completion.